CLINICAL TRIAL: NCT06609395
Title: Pilot Study Testing an Online-delivered Psychological Intervention for Indian Expatriates in Sweden Who Experience Dysfunctional Worry
Brief Title: Brief Online Cognitive Behavioral Therapy for Indian Expatriates with Excessive Worry: a Pilot Feasibility Study
Acronym: Worry-exp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Nitya Jayaram-Lindstrom, PhD, Director of Centre for Psychiatry Research, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Worry-exp; 000 (Other Grant/Funding Number: RaD grants, Stockholm Health Care Services, Region Stockholm)
Record Dates: First submitted 2024-09-22; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Excessive Worry
Keywords: Digital CBT, Brief intervention, Indian Expatriate

STUDY DESIGN:
Intervention Model Description: Open pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brief online CBT targeting excessive worry (Experimental): The treatment in this trial was based on an online CBT intervention developed by Wahlund et al. (2021) for dysfunctional worry during the COVID-19 pandemic. Originally designed for the Swedish population, the intervention was translated to English and adapted for Indian expatriates in Sweden, addressing broader global crises, including military conflicts and climate change.
  Interventions: Behavioral: Brief online CBT targeting excessiv worry

INTERVENTIONS:
Behavioral: Brief online CBT targeting excessiv worry — The intervention with a focus on excessive worry lasted five weeks and was delivered through five online modules with therapist support. Modules covered psychoeducation, problem-solving, reducing excessive media consumption, detached mindfulness, and shifting focus from worry. The final module offered relapse prevention strategies.

SUMMARY:
Background: Expatriates may face challenges through distance from support systems, cultural adjustments, and language barriers, which may be associated with anxiety and elevated worry, particularly in times of ongoing global crises. Brief online cognitive-behavioral therapy (ICBT) is effective for treating excessive worry but has not been adapted for expatriate communities in Sweden.

DETAILED DESCRIPTION:
This pilot study aimed to investigate the feasibility, acceptability, and preliminary treatment effects of a five-week, therapist-guided, culturally adapted ICBT program. The program targeted excessive worry related to ongoing global crises among Indian expatriates.

ELIGIBILITY:
Inclusion Criteria:

* identifying as Indian expatriate currently living in Sweden
* self-reported dysfunctional worry, defined as worrying several times a day and the worry being experienced as difficult to control
* age ≥ 18 years;
* able to provide digital informed consent
* having daily access to a device with internet connection.

Exclusion Criteria:

* non-English speaking
* self-reported severe depression (>28 points on the Montgomery Åsberg Depression Rating Scale (MADRS-S; (Svanborg & Åsberg, 1994)
* suicidal risk (5 points on item 9 on the MADRS-S).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder Scale-7 (GAD-7) | Baseline to post-treatment (5 weeks)
  The GAD-7 is a 7-item self-report tool used to assess generalized anxiety disorder severity. It scores symptoms like worry and restlessness over the past two weeks on a scale of 0 to 3, with a total score of 0-21. Scores categorize anxiety as mild, moderate, or severe.
Generalized Anxiety Disorder Scale-7 (GAD-7) | Baseline to 1-month follow-up ( 9 weeks)
  The GAD-7 is a 7-item self-report tool used to assess generalized anxiety disorder severity. It scores symptoms like worry and restlessness over the past two weeks on a scale of 0 to 3, with a total score of 0-21. Scores categorize anxiety as mild, moderate, or severe.

SECONDARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale - Self report (MADRS-S) | Baseline to post-treatment (5 weeks)
  The MADRS-S is a 9-item self-report scale for assessing depression severity. Each item is scored 0 to 6, with higher scores reflecting more severe symptoms like mood, sleep, and concentration issues.
Montgomery Åsberg Depression Rating Scale - Self report (MADRS-S) | Baseline to 1-month follow-up ( 9 weeks)
  The MADRS-S is a 9-item self-report scale for assessing depression severity. Each item is scored 0 to 6, with higher scores reflecting more severe symptoms like mood, sleep, and concentration issues.
Work and Social Adjustment Scale (WSAS) | Baseline to post-treatment (5 weeks)
  The WSAS is a 5-item self-report scale measuring how mental health issues affect work, home tasks, social life, and relationships. Higher scores indicate greater impairment.
Work and Social Adjustment Scale (WSAS) | Baseline to 1-month follow-up ( 9 weeks)
  The WSAS is a 5-item self-report scale measuring how mental health issues affect work, home tasks, social life, and relationships. Higher scores indicate greater impairment.
Insomnia Severity Index | Baseline to post-treatment (5 weeks)
  The Insomnia Severity Index (ISI) is a 7-item scale assessing insomnia severity, including sleep issues and daytime impact. Higher scores indicate more severe insomnia.
Insomnia Severity Index | Baseline to 1-month follow-up ( 9 weeks)
  The Insomnia Severity Index (ISI) is a 7-item scale assessing insomnia severity, including sleep issues and daytime impact. Higher scores indicate more severe insomnia.
Client Satisfaction Questionnaire CSQ | Baseline to post-treatment (5 weeks)
  The Patient Satisfaction Questionnaire (PSQ) is a self-report tool that measures patients' satisfaction with healthcare services. It covers aspects like quality of care, communication, convenience, and overall experience. Higher scores indicate greater satisfaction.
  The Patient Satisfaction Questionnaire (PSQ) is a self-report tool that measures patients' satisfaction with intervention. It covers aspects like quality of care, communication, convenience, and overall experience. Higher scores indicate greater satisfaction.
  he Patient Satisfaction Questionnaire (PSQ) measures patients' satisfaction with healthcare, focusing on care quality, communication, and convenience. Higher scores show greater satisfaction.
Adverse events | Baseline to post-treatment (5 weeks)
  Adverse events for participating in the intervention may include increased anxiety, emotional distress, or frustration. Patients rate the severity and duration of these events on a scale from 0 to 3.
Adverse events | Baseline to 1-month follow-up ( 9 weeks)
  Adverse events for participating in the intervention may include increased anxiety, emotional distress, or frustration. Patients rate the severity and duration of these events on a scale from 0 to 3.
Adherence to treatment | From baseline to treatment (5 weeks)
  Treatment completion was defined as a participant successfully finishing at least four out of the five treatment modules (described below) included returning the associated homework assignment linked to each module. This level was set as modules 1-4 provide the core components of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nitya Jayaram-Lindström, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Centre for Psychiatry Research, Karolinska Institutet, Stockholm Healthcare Services, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
GDPR is not allowing.

REFERENCES:
- [Background] Uvais NA, Nalakath MJ, Shihabudheen P, Hafi NAB, Salman CA. Depression, Anxiety, and Coping During the COVID-19 Pandemic Among Indian Expats in the Middle East: A Survey Study. Prim Care Companion CNS Disord. 2021 Jan 21;23(1):20m02761. doi: 10.4088/PCC.20m02761. PMID 33480484
- [Background] Vijayakumar, P. B., & Cunningham, C. J. L. (2016). Cross-cultural adjustment and expatriation motives among Indian expatriates. Journal of Global Mobility: The Home of Expatriate Management Research, 4(3), 326-344. https://doi.org/10.1108/jgm-05-2016-0019
- [Background] Zhou ES, Ritterband LM, Bethea TN, Robles YP, Heeren TC, Rosenberg L. Effect of Culturally Tailored, Internet-Delivered Cognitive Behavioral Therapy for Insomnia in Black Women: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Jun 1;79(6):538-549. doi: 10.1001/jamapsychiatry.2022.0653. PMID 35442432
- [Background] Wahlund T, Mataix-Cols D, Olofsdotter Lauri K, de Schipper E, Ljotsson B, Aspvall K, Andersson E. Brief Online Cognitive Behavioural Intervention for Dysfunctional Worry Related to the COVID-19 Pandemic: A Randomised Controlled Trial. Psychother Psychosom. 2021;90(3):191-199. doi: 10.1159/000512843. Epub 2020 Nov 19. PMID 33212440